CLINICAL TRIAL: NCT03549507
Title: Evaluation of Bowel Perfusion With Contrast-Enhanced Ultrasound in Necrotizing Enterocolitis
Brief Title: CEUS Evaluation of Bowel Perfusion in Necrotizing Enterocolitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Bracco Diagnostics, Inc (Industry)
Responsible Party: Principal Investigator, Misun Hwang, MD, Sponsor Investigator, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-014910
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Necrotizing Enterocolitis of Newborn; Bowel Ischemic
Keywords: Ultrasound; Contrast-enhanced ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Contrast-enhanced Ultrasonography (Experimental): Intravenous administration of contrast agent Sulfur hexafluoride lipid-type A microspheres before performing contrast-enhanced ultrasound (CEUS). In pediatric patients, after reconstitution 0.03 mL per kg is administered intravenously. The weight-based dose of 0.03 mL per kg will be repeated one time during a single examination. Following each injection, an intravenous flush of 0.9% Sodium Chloride is injected. The study duration per subject will be approximately 15 minutes including the time to prepare the contrast agent and perform the CEUS, as well as the 60 minute monitoring period after the first and second injection (if there are two injections of contrast) of the contrast agent.
  Interventions: Drug: Sulfur hexafluoride lipid-type A microspheres

INTERVENTIONS:
Drug: Sulfur hexafluoride lipid-type A microspheres — Injection of Sulfur hexafluoride lipid-type A microspheres (Lumason) contrast agent will be performed via the existing peripheral intravenous line using the FDA-recommended dose of 0.03 mg/kg. Two bolus injections will be performed to evaluate for dynamic bowel perfusion and several 2-minute cine clips as well as static images will be acquired during the exam.

SUMMARY:
There is no bedside imaging technique that can quantify dynamic bowel perfusion with high soft tissue contrast and sensitivity in necrotizing enterocolitis (NEC). Our goal is to assess the feasibility of utilizing contrast-enhanced ultrasound (CEUS) in bedside monitoring of bowel perfusion in NEC. Patients with suspected or diagnosed NEC will be recruited for the study. Following parental consent, the subject will undergo CEUS, performed separately from any clinically indicated conventional US, in the ICU. Subjects will be scanned with CEUS at two different time-points (at the time NEC is first suspected or diagnosed and at time of MRI scan). The CEUS scans will be interpreted by the sponsor-investigator.

The study will be conducted at one site, The Children's Hospital of Philadelphia. It is expected that up to 100 subjects will be enrolled per year, for up to two years, for a total enrollment of up to 200 subjects.

DETAILED DESCRIPTION:
Early detection of ischemia and necrotic bowel which leads to perforation is vital in improving morbidity and mortality associated with NEC. Abdominal radiography, the standard imaging algorithm for monitoring of NEC, has a low sensitivity of 40% in the diagnosis of severe NEC with necrotic bowel. There is a dire need to introduce better imaging tools such as CEUS to the clinical setting that can detect NEC at an early stage and prompt therapeutic implementation. CEUS enables safe, serial monitoring of dynamic quantification of bowel perfusion at the bedside.

Sulfur hexafluoride lipid-type A microspheres (LumasonTM, Bracco Inc) is an FDA-approved ultrasound contrast agent. The study duration per subject will be approximately 15 minutes including the time to prepare LumasonTM contrast agent and perform the CEUS, as well as the 60 minute monitoring period after the first and second injection of LumasonTM. CEUS will be performed at the time of suspected or diagnosed NEC, and at the time of surgery (for subjects undergoing surgery as part of clinical care) or at short-term follow-up of clinical condition (approximately 1 week after the first scan) for a total of two CEUS exams of 1 hour and 15-minute duration each.

Injection of LumasonTM contrast agent will be performed via the existing peripheral intravenous line or central line using the FDA-recommended dose of up to 0.03 mg/kg. Contrast-agent injection will be performed twice per CEUS scan to ensure image quality and test reproducibility. In the case of more stable patients without an IV line, a peripheral IV line will be started to conduct the investigational CEUS. Two bolus injections will performed to evaluate for dynamic bowel perfusion and several 2-minute cine clips as well as static images will be acquired during the exam.

Qualitative analysis with visual assessment and quantitative analysis of the acquired CEUS scans will be performed and interpreted by the PI. The scans will be assessed for diagnostic quality of images, artifacts encountered, and the presence of additional contributory diagnostic information.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 1.5 years or younger
2. Post menstrual age of 29 weeks or older
3. Patients with suspected or diagnosed necrotizing enterocolitis
4. Patient in the Children's Hospital of Philadelphia (CHOP) neonatal intensive care unit (NICU) or pediatric intensive care unit (PICU)
5. Parental permission

Exclusion Criteria:

1. Medical history of Lumason hypersensitivity
2. Hemodynamic instability as defined by rapid escalation of cardiopulmonary support in the past 12-24 hours, as defined by the clinical care team including ≥ 1 intensive care physician not part of the study team
3. Pulmonary insufficiency as defined by FiO2 requirements of >40% and/or subjects with pulmonary hypertension requiring nitric oxide

Ages: 0 Years to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Misun Hwang, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang M, Piskunowicz M, Darge K. Advanced Ultrasound Techniques for Pediatric Imaging. Pediatrics. 2019 Mar;143(3):e20182609. doi: 10.1542/peds.2018-2609. PMID 30808770

RESULTS

PARTICIPANT FLOW:
Groups:
- Bowel Contrast-enhanced Ultrasonography: Intravenous administration of contrast agent Sulfur hexafluoride lipid-type A microspheres before performing contrast-enhanced ultrasound (CEUS). In pediatric patients, after reconstitution 0.03 mL per kg is administered intravenously. The weight-based dose of 0.03 mL per kg will be repeated one time during a single examination. Following each injection, an intravenous flush of 0.9% Sodium Chloride is injected. The study duration per subject will be approximately 15 minutes including the time to prepare the contrast agent and perform the CEUS, as well as the 60 minute monitoring period after the first and second injection (if there are two injections of contrast) of the contrast agent.
  Sulfur hexafluoride lipid-type A microspheres: Injection of Sulfur hexafluoride lipid-type A microspheres (Lumason) contrast agent will be performed via the existing peripheral intravenous line using the FDA-recommended dose of 0.03 mg/kg. Two bolus injections will be performed to evaluate for dynamic bowel perfusion and several 2-minute cine clips as well as static images will be acquired during the exam.
Period: Overall Study
Arm/Group | Bowel Contrast-enhanced Ultrasonography
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Low enrollment. Main reason was not fulfillment of inclusion/exclusion criteria, either for clinical instability and/or pulmonary insufficiency/hypertension.
Arm/Group | Contrast-enhanced Ultrasonography
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 47 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Early Detection of Altered Bowel Perfusion Using CEUS
Description: Comparison of bowel perfusion between normal subjects (those with suspected or at risk of necrotizing enterocolitis but turn out to be normal on imaging and clinical evaluation) versus NEC patients
Time Frame: 2 years
Population: One subject was enrolled, therefore, no comparison was possible. The enrolled subject presented with medical NEC. Main reasons for lack of enrollment were the presence of clinical instability and/or pulmonary insufficiency/hypertension.
Measure: Number; unit: Number of patients
Groups:
- Bowel Contrast-enhanced Ultrasonography: Intravenous administration of contrast agent Sulfur hexafluoride lipid-type A microspheres before performing CEUS through an existing peripheral intravenous line using the FDA-recommended dose of 0.03 mg/kg. Two bolus injections will be performed and several 2-minute cine clips as well as static images will be acquired during the exam.
Arm/Group | Bowel Contrast-enhanced Ultrasonography
Number analyzed (Participants) | 1
Number of patients
  Patients with NEC who underwent CEUS examination | 1
  Patients without NEC who underwent CEUS examination | 0

2. Secondary Outcome: Number of Participants With Completed CEUS Exams, Categorized by Diagnostic-Quality Scoring System
Description: Scoring system of non-diagnostic (1), moderate artifacts degrading diagnostic quality (2), mild artifacts without degradation of diagnostic quality (3), and diagnostic (4).
Time Frame: 2 years
Population: Evaluation of CEUS diagnostic quality
Measure: Number; unit: Number of participants
Arm/Group | Bowel Contrast-enhanced Ultrasonography
Number analyzed (Participants) | 1
Number of participants
  Non-diagnostic | 0
  Mild artifacts without degradation of diagnostic quality | 0
  Moderate artifacts degrading diagnostic quality | 1
  Diagnostic | 0

ADVERSE EVENTS:
Time Frame: 15 Minutes.
Arm/Group | Bowel Contrast-enhanced Ultrasonography
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT03549507/Prot_SAP_000.pdf